CLINICAL TRIAL: NCT00751647
Title: Cystic Fibrosis Core Strengthening and Respiratory Exercise Program (CSREP)
Brief Title: Cystic Fibrosis Core Strengthening and Respiratory Exercise Program
Acronym: CSREP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0807-068
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Cystic Fibrosis
Keywords: CF
MeSH Terms: conditions — Cystic Fibrosis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A1 (Other): Population receiving the CF specific outpatient PT services.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — Treatment

SUMMARY:
The purpose of this project is to determine the short-term effects of a customized Core Strengthening and Respiratory Exercise Program (CSREP) on children with cystic fibrosis (CF) between the ages of 10 and 21 who are receiving outpatient care at Children's Hospitals and Clinics of Minnesota. The CSREP, which will be provided by a physical therapist and a physical therapist assistant, consists of specific breathing techniques and core strengthening exercises, designed to improve rib cage mobility, pulmonary function, aerobic capacity, posture, and core strength. Currently the CF population at Children's receives physical therapy on an inpatient basis only.

The overall goal of this program is to prove the viability of an outpatient exercise program for this population. Specific aims include:

* To customize a CSREP protocol per each patient
* To measure patient outcomes at baseline and six months
* To develop a satisfaction tool in order to measure patient experience and satisfaction

DETAILED DESCRIPTION:
Study Design: Phase II clinical trial.

Objective: To determine whether a customized physical therapy exercise intervention titled Core Strengthening and Respiratory Exercise Program (CSREP) clinically improves the following outcome measures for children between the ages of 10 and 21 with cystic fibrosis: pulmonary function, aerobic capacity, rib cage mobility, posture, and core strength, thus warranting more extensive study and development.

Background: Previous research conducted in pediatric populations has focused on the effects of aerobic training, anaerobic training, and strengthening of the extremities on the health of children with cystic fibrosis. However, the disease process of cystic fibrosis secondarily causes impairments in the musculoskeletal and nervous systems. No intervention study aimed at positively impacting these systems has been done to date with children with cystic fibrosis.

Methods: A 6-month CSREP will be customized to meet the specific needs of each participant. During Part I of the program participants will attend weekly CSREP treatments for 4 to 6 weeks; in Part II they will attend monthly CSREP treatments over a five-month period. Each session will last for 45-60 minutes. During these treatments, participants will be given instruction on a daily home exercise program and will receive hands on physical therapy interventions. Handouts with pictures and how-to instructions for assigned exercises will be provided. Participants will be given calendars to track completion of home exercises and level of compliance. During Part II, a researcher will call participants every week in order to encourage compliance with the home exercise program and to provide clarification as needed. All participants will continue to receive regular medical care as well as PT treatments.

A respiratory therapist will perform the pulmonary function tests, a respiratory therapist along with an exercise physiologist will perform the VO2max testing, and a physical therapist will perform the physical therapy evaluation, including assessment of rib cage mobility, core strength, and posture. Another physical therapist as well as a physical therapist assistant will provide the physical therapy treatments, instruct the participants in their home program, and make the weekly phone calls to all participants.

An experience survey will be designed to evaluate both satisfaction on a scale of 1 to 10 and self scoring of outcome measures including: respiratory function, cough strength, activity tolerance, posture, and strength on a three point Likert scale of: 1) Got worse; 2) Stayed the same; and 3) Got better. Additionally, the survey will include a question on the likelihood of continuing with the home program after the study has ended. The survey will be administered at 6 months upon completion of the program.

Relevance: The results of this inquiry as to the viability of the CSREP will prove relevant to the above-mentioned patient outcomes within the cystic fibrosis population. The customized CSREP protocol will provide a non-pharmacological outpatient treatment option that can be completed on an outpatient basis, independently, in the patient's home.

ELIGIBILITY:
Inclusion criteria:

* Children with cystic fibrosis receiving outpatient care from Children's Cystic Fibrosis Clinic
* Aged 10-21
* Living within a 35-mile radius of Children's Minneapolis, who agree to participate.

Exclusion Criteria:

* Children with co-morbid conditions in which the exercise program is contra-indicated will be excluded from this study.

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2008-12; Primary Completion 2012-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Pulmonary function, aerobic capacity, rib cage mobility, posture, and core strength, thus warranting more extensive study and development. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Katie Fenlon, PT, Principal Investigator — Children's Hospitals and Clinics of MN
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota, United States